CLINICAL TRIAL: NCT03014206
Title: PREVENAR13(REGISTRIED) SUSPENSION LIQUID FOR INJECTION DRUG USE INVESTIGATION - ADULTS AGED 65 YEARS OR OLDER
Brief Title: Prevenar13 Drug Use Investigation - Adults Aged 65 Years or Older-
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: B1851121
Record Dates: First submitted 2016-07-18; First posted 2017-01-09 (Estimated); Results first posted 2019-02-28 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-08

CONDITIONS: Adult Not Younger Than 65 Years

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 28 Days
Oversight: Data Monitoring Committee: No

SUMMARY:
This study aims to understand the following items in post-marketing actual clinical settings to evaluate the safety of 13vPnC administered as a single dose in the elderly (adults aged 65 years or older).

1. To confirm the use in actual clinical settings
2. To confirm the occurrence of adverse events

DETAILED DESCRIPTION:
This study is a multicenter open-label cohort conducted in patients vaccinated with the Product; for which, case report forms will be recorded based on data presented in medical records obtained from day-to-day clinical treatment and diagnosis. "Pneumococcal vaccine health study diary" will be implemented to collect accurate safety data; to which, vaccine recipients will be asked directly to cooperate.

ELIGIBILITY:
Inclusion Criteria:

1. Geriatric patients vaccinated with this product (adult not younger than 65 years)
2. Consent of vaccine recipients [Vaccine recipient (or his/her legally acceptable representative) must sign and date the consent form warranting that the relevant information concerning this Study was appropriately communicated to the recipient].

Exclusion Criteria:

None

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Geriatric patients vaccinated with this product (adult not younger than 65 years)
Sampling Method: Probability Sample
Enrollment: 696 (Actual)
Dates: Start 2015-06-15 (Actual); Primary Completion 2017-01-31 (Actual); Study Completion 2017-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1851121&StudyName=Prevenar%20%2813v%29%20Adult%20Special%20Investigation%20%28regulatory%20Post%20Marketing%20Commitment%20Plan%29

RESULTS

PARTICIPANT FLOW:
Groups:
- Prevenar 13 (Pneumococcal 13-valent Conjugate Vaccine): Participants who received Prevenar 13 as indicated in the approved local product document were observed for a period of 28 days.
Period: Overall Study
Arm/Group | Prevenar 13 (Pneumococcal 13-valent Conjugate Vaccine)
Started | 696
Completed | 684
Not Completed | 12
Not completed — Registration Violation | 12

BASELINE CHARACTERISTICS:
Population: A total of 696 participants were enrolled in this study. Of the 696 participants, 12 participants were excluded from the baseline analysis due to registration violation.
Arm/Group | Prevenar 13 (Pneumococcal 13-valent Conjugate Vaccine)
Number analyzed (Participants) | 684
Age, Customized [Number; unit: Participants]
  <65 years | 0
  ≥65 and <70 years | 127
  ≥70 and <75 years | 157
  ≥75 and <80 years | 154
  ≥80 and <85 years | 134
  ≥85 years | 112
Sex/Gender, Customized [Number; unit: Participants]
  Female | 385
  Male | 299
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 684

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Reactions
Description: An adverse reaction (vaccine-related adverse event) was any untoward medical occurrence attributed to Prevenar 13 in a participant who received Prevenar 13. A serious adverse reaction was a vaccine-related adverse event resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Relatedness to Prevenar 13 was assessed by the physician.
Time Frame: 28 days
Population: The safety analysis set comprised of participants who satisfied the inclusion criteria and provided the safety data after vaccination with Prevenar 13.
Measure: Number; unit: Participants
Arm/Group | Prevenar 13 (Pneumococcal 13-valent Conjugate Vaccine)
Number analyzed (Participants) | 684
Participants
  Adverse Reactions | 80
  Serious Adverse Reactions | 1

ADVERSE EVENTS:
Time Frame: 28 days
Description: The frequency of adverse events. The same event may appear as both an adverse event and a serious adverse event. However, what is presented are distinct events. An event may be categorized as serious in one subject and as non-serious in another subject, or one subject may have experienced both serious and non-serious events during the study.
Arm/Group | Prevenar 13 (Pneumococcal 13-valent Conjugate Vaccine)
All-Cause Mortality (participants affected / at risk) | 0/684
Serious Adverse Events (participants affected / at risk) | 6/684
Other Adverse Events (participants affected / at risk) | 85/684
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prevenar 13 (Pneumococcal 13-valent Conjugate Vaccine) (N=684)
Pneumonia (Infections and infestations) | 1 (1)
Vaccination site cellulitis (Infections and infestations) | 1 (1)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Prevenar 13 (Pneumococcal 13-valent Conjugate Vaccine) (N=684)
Nausea (Gastrointestinal disorders) | 1
Injection site hypoaesthesia (General disorders) | 1
Malaise (General disorders) | 2
Pneumonia (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Vaccination complication (Injury, poisoning and procedural complications) | 1
Blood creatine phosphokinase increased (Investigations) | 1
Rash generalised (Skin and subcutaneous tissue disorders) | 1
Pyrexia (General disorders) | 10
Vaccination site dermatitis (General disorders) | 1
Vaccination site erythema (General disorders) | 35
Vaccination site pain (General disorders) | 34
Vaccination site pruritus (General disorders) | 6
Vaccination site swelling (General disorders) | 36

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2016-07-22): https://cdn.clinicaltrials.gov/large-docs/06/NCT03014206/Prot_001.pdf
  • Statistical Analysis Plan (2016-12-08): https://cdn.clinicaltrials.gov/large-docs/06/NCT03014206/SAP_000.pdf